CLINICAL TRIAL: NCT01638065
Title: A Comprehensive Look at Vascular Access: Utilizing a Near Infrared Vein Visualization Device For Vascular Access Planning, Attempts, and Post Access
Brief Title: A Comprehensive Look at Vascular Access
Status: Completed | Type: Observational
Sponsor: Christie Medical Holdings, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP1011
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Vascular Access
Keywords: vein identification; vascular access

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard: Standard IV Access without device
- VeinViewer: IV access with VeinViewer device

SUMMARY:
The objective of this study is to show VeinViewer® Vision is an effective vein visualization device for peripheral vascular access, pre-, during, and post access.

ELIGIBILITY:
Inclusion Criteria:

* Requires peripheral venous access
* Intact skin on areas of assessment
* Patient and/or parent or legal guardian is able to understand consent

Exclusion Criteria:

* No Intact skin
* Patient is under anesthesia during peripheral venous access
* Patient is not a suitable candidate, as determined by the discretion of the investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at a medical facility requiring IV access.
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be total number of attempts for successful cannulation. | 1 day

SECONDARY OUTCOMES:
Amount of time for successful venous access | 1 day

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - LA County Hospital, Los Angeles, California
  - Good Samaritan Hospital, Downers Grove, Illinois